CLINICAL TRIAL: NCT03947762
Title: Lanreotide 120 mg Effectiveness in Subjects With Locally Advanced or Metastatic Pancreatic Neuroendocrine Tumours (PanNET) in Routine Clinical Practice
Brief Title: Lanreotide 120mg Effectiveness in Subjects With Pancreatic Neuroendocrine Tumours (PanNET) in Routine Clinical Practice.
Acronym: PanNET
Status: Terminated | Type: Observational
Why Stopped: Low enrollment
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-ES-52030-383; IPS-LAN-2018-01 (Other: Spanish Drug Agency AEMPS)
Record Dates: First submitted 2019-05-10; First posted 2019-05-13 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Pancreatic Neuroendocrine Tumor
MeSH Terms: conditions — Adenoma, Islet Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the protocol is to estimate the progression-free survival (PFS) rate in subjects diagnosed with PanNET, according to investigator assessment, at 24 months after treatment initiation with lanreotide 120 mg every 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥ 18
* Subjects diagnosed of functioning or non-functioning PanNET, G1/ G2 (Ki67≤10%) unresectable locally advanced tumour or metastatic disease, who have been treated with lanreotide 120mg every 28 days for at least 3 months and a maximum of 12 months
* Subject not progressive at inclusion study visit according to investigator assessment, and using as a reference lanreotide initiation
* Subject with Eastern Cooperative Oncology Group (ECOG) ≤2

Exclusion Criteria:

* Subject who is participating in an interventional study
* Pregnant or breast-feeding women
* Subject who has received any previous therapy for PanNET (such as octreotide LAR, Molecular Targeted Therapy (MTT), Peptide receptor radionuclide therapy (PRRT), chemotherapy, etc.) except short-acting octreotide subcutaneous (SC) used for symptomatic control of functioning tumours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital patients
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate at 24 months | 24 months
  To estimate the progression-free survival (PFS) rate in subjects diagnosed with PanNET, according to investigator assessment.

SECONDARY OUTCOMES:
Progression-free survival (PFS) rate at 12 months | 12 months
  PFS rate at 12 months after lanreotide treatment initiation according to investigator assessment
Medical tumour-related intervention | Baseline
  Description of the disease history management of subjects with PanNET will be collected by the investigator and recorded in an electronic CRF (eCRF) designed for the study
Time from diagnosis to first therapeutic intervention | Baseline
  Description of the disease history management of subjects with PanNET
Quality of Life (QoL) | From baseline up to 24 months
  To describe the change in Quality of Life (QoL) as assessed by European Organisation for Research and Treatment of Cancer (EORTC) QoL questionnaire for gastrointestinal neuroendocrine tumours (QLQ-GINET21) questionnaires.Where the patient assess experienced symptoms or problems using the scale from 1 to 4. Where 1 represents "not at all" and 4 "very much".
Median time to lanreotide discontinuation | Up to 24 months
Changes of Chromogranin A (CgA) levels | Every 6 months up to 24 months
  Changes in CgA levels between last CgA value prior to lanreotide start (if available) and values at each study visit
Changes of Glycated hemoglobin (HbA1c) levels | Every 6 months up to 24 months
  Changes in HbA1c levels between last HbA1c value prior to lanreotide start (if available) and values at each study visit
Changes of urine 5-Hydroxyindoleacetic Acid (5-HIAA) levels | Every 6 months up to 24 months
  Changes in 5-HIAA levels between last 5-HIAA value prior to lanreotide start (if available) and values at each study visit
Changes of pro-Brain Natriuretic Peptide (proBNP) levels | Every 6 months up to 24 months
  Changes in proBNP levels between last proBNP value prior to lanreotide start (if available) and values at each study visit
Patient satisfaction | Baseline visit and 12 months
  To evaluate patient' satisfaction (TSQM-9 questionnaire) at inclusion visit. Treatment Satisfaction Questionnaire for Medication (TSQM) is an instrument to assess patients' satisfaction with medication, providing scores on four scales - side effects, effectiveness, convenience and global satisfaction. The effectiveness scored as: 1 (extremely dissatisfied) to 7 (extremely satisfied). For the convenience scored as 1(extremely difficult) to 7 (extremely easy).

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (46):
- Portugal (3):
  - IPO Coimbra, Coimbra
  - IPO Lisboa, Lisbon
  - Hospital São João, Porto
- Spain (43):
  - Hospital General de Alicante, Alicante
  - Hospital Torrecardenas, Almería
  - Hospital Universitario de Badajoz, Badajoz
  - ICO Badalona, Badalona
  - Hospital de Cruces, Barakaldo
  - Hospital Universitario Vall Hebrón, Barcelona
  - Hospital Santa Creu I Sant Pau, Barcelona
  - Hospital Basurto, Bilbao
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Puerto Real, Cadiz
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital General Ciudad Real, Ciudad Real
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Donostia, Donostia / San Sebastian
  - Hospital Virgen de las Nieves, Granada
  - Hospital Juan Ramón Jimenez, Huelva
  - Hospital Can Misses, Ibiza Town
  - Hospital de Jerez, Jerez de la Frontera
  - ICO Bellvitge, L'Hospitalet de Llobregat
  - Hospital U. de Gran Canaria Negrín, Las Palmas de Gran Canaria
  - Hospital Virgen de La Victoria, Málaga
  - Hospital Clínico U. Virgen de la Arrixaca, Murcia
  - Hospital Morales Meseguer, Murcia
  - Hospital Santa María Nai, Ourense
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Son Espases, Palma de Mallorca
  - Hospital de Navarra, Pamplona
  - Hospital Sant Joan de Reus, Reus
  - Corporació Sanitària Parc Taulí, Sabadell
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital U. Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Hospital Marqués de Valdecillas, Santander
  - Hospital Conxo, Santiago de Compostela
  - Hospital General de Segovia, Segovia
  - Hospital Virgen Macarena, Seville
  - Hs. Virgen del Rocio, Seville
  - Hospital Mutua Terrassa, Terrassa
  - Hospital Virgen de la Salud Toledo, Toledo
  - Hospital General de Valencia, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Álvaro Cunqueiro, Vigo
  - Hospital Lozano Blesa, Zaragoza
  - Hospital Miguel Servet, Zaragoza